CLINICAL TRIAL: NCT05207514
Title: Open-label, Randomized, Active-controlled, Multicenter, Phase III Clinical Trial to Compare the Efficacy and the Safety of Taxotere and Nanoxel M as Neoadjuvant Chemotherapy in Breast Cancer
Brief Title: Compare the Efficacy and the Safety of Taxotere and Nanoxel M as Neoadjuvant Chemotherapy in Breast Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The Decision to Terminate Early Due to Difficulties in Recruiting Participants and Conducting the Study.
Sponsor: Samyang Biopharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DPMBC301
Record Dates: First submitted 2022-01-07; First posted 2022-01-26 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Polysorbates; Docetaxel; Doxorubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nanoxel M (Experimental): AC(Doxorubicin, Cyclophosphamide) followed by Nanoxel M
  Interventions: Drug: Nanoxel M; Drug: Doxorubicin; Drug: Cyclophosphamide
- Taxotere (Active Comparator): AC(Doxorubicin, Cyclophosphamide) followed by Taxotere
  Interventions: Drug: Taxotere; Drug: Doxorubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Nanoxel M — 75 mg/m2, intravenously every 3 weeks for 4 cycles (after treatment cycles of doxorubicin and cyclophosphamide
  Other Names: polysorbate 80, ethanol free docetaxel
  Arms: Nanoxel M
Drug: Taxotere — 75 mg/m2, intravenously every 3 weeks for 4 cycles (after treatment cycles of doxorubicin and cyclophosphamide
  Other Names: docetaxel
  Arms: Taxotere
Drug: Doxorubicin — 60 mg/m2, intravenously every 3 weeks for 4 cycles. Given as first treatment with cyclophosphamide
Drug: Cyclophosphamide — 600 mg/m2, intravenously every 3 weeks for 4 cycles. Given as first treatment with doxorubicin.

SUMMARY:
Phase III Clinical Trial to Compare the Efficacy and the Safety of AC(Doxorubicin, Cyclophosphamide) Followed by 4 Cycles Taxotere Versus AC(Doxorubicin, Cyclophosphamide) Followed by 4 Cycles Nanoxel M as Neoadjuvant Chemotherapy in Patients With Breast Cancer

DETAILED DESCRIPTION:
The purpose of this study is to evaluate efficacy and safety of AC followed by Taxotere versus AC followed by Nanoxel M as neoadjuvant chemotherapy in breast caner patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who were diagnosed with primary breast cancer by core biopsy
2. Patients who have been identified as HER2 negative in the tissue obtained through core needle biopsy and have confirmed the positive / negative status of ER (Estrogen receptor) and Progesterone receptor (PR)

   * HER2 positive is defined as IHC 3+ or FISH +
3. Patinets whose TNM stage confirmed by CT or MRI (T2-T3, anyN, M0 or T1-3, N1-3, M0)

Exclusion criteria:

1. Patients who have distant metastasis
2. Patients who have cystitis or urinary obstruction
3. Patients who have history of thromboembolism or coagulation disorder
4. Patients who have Interstitial lung disease ans liver cirrhosis ( > Child-Pugh class B)
5. Patients who have Insulin-Dependent Type II diabete mellitus

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-05-09 (Actual)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate using the definition of ypT0/Tis ypN0 | at the time of definitive surgery
  H & E staining of tissues obtained from breast and axillary lymph nodes was defined as the absence of invasive cancer, and the proportion of subjects was determined.

CONTACTS AND LOCATIONS:
Overall Officials: Joohyuk Sohn, M.D.,Ph.D., Principal Investigator — Severance Hospital
Locations (1):
- Sevrance Hospital, Seoul, South Korea